CLINICAL TRIAL: NCT05020054
Title: Effect of Tecartherapy in the Treatment of Localized Fat and Sagging Abdominal Skin - Clinical and Experimental Study
Acronym: Tecarterapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Tecarterapy
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Fat Disorder; Fat Redistribution
Keywords: fat disorder; fat redistribution
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: tecarterapia intervention and placebo
Who Masked: Participant
Masking Description: the participant did not know that the therapy was placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Tecartherapy (Active Comparator): The procedures will be performed with Tecartherapy equipment, with the equipment Nèartek®- IBRAMED- Industria Brasileira de Equipamentos Eletromédicos.
  The treatment will be carried out once a week, totaling 10 sessions, by two dermato-functional physiotherapists. During the sessions, all volunteers will be positioned in dorsal decubitus and the applicator positioned in the abdominal region, the therapy will be dynamic and simultaneously the professional must assess the local temperature.
  The parameters used will be:
  Area of 300cm², 1MHz, Capacitive Mode: 60mm Disc: Default 100W Time of 10 minutes, keeping temperature at 42°C Resistive Mode: 60mm Disc: Default 110W Time of 10 minutes, keeping temperature at 42ºC. The total treatment time is 20 minutes.
  Interventions: Device: Tecartherapy Intervention
- Placebo Tecartherapy (Placebo Comparator): the therapy took place with the equipment turned off
  Interventions: Device: placebo tecartherapy

INTERVENTIONS:
Device: Tecartherapy Intervention — therapeutic therapy with effective application, connected equipment
  Other Names: Intervention
  Arms: Intervention Tecartherapy
Device: placebo tecartherapy — tecartherapy with equipment turned off
  Arms: Placebo Tecartherapy

SUMMARY:
The excess of localized fat causes changes in the body contour and consequently changes in the properties of the skin and in the connective tissue, providing sagging skin.

Tecartherapy known as High Frequency Capacitive and Resistive Electrical Transfer Therapy (Tecartherapy) emerged to contribute to the treatment of these aesthetic affections, it is a non-invasive electrothermal therapy that acts on cell biostimulation through tissue heating and can help to reduce fat localized and improve the aspect of flaccidity, through the stimulation of neocollagenesis and neoelastogenesis.

This is the aim of this research is to evaluate the effects of Tecartherapy on localized fat and abdominal skin flaccidity with clinical and histological results.

The sample will have 61 participants, who will be evaluated pre and post treatment through evaluation protocols, photographs and questionnaires. The research will have two treatment groups. Being Group 1: Tecartherapy and Group 2: placebo (equipment turned off). 10 Tecartherapy sessions will be held once a week in the abdominal region and flanks. The parameters used will be: for an area of 300cm², 1MHz, Capacitive Mode: 60mm Disk, Default 100W, Time of 10 minutes, keeping temperature up to 42ºC, Resistive Mode: 60mm Disk: Default 110W, Time of 10 minutes, keeping temperature up to 42ºC, with a total treatment time of 20 minutes for the 300cm² area.

After treatment, a biopsy of the subcutaneous tissue and skin will be performed in a volunteer, the tissue will be collected during the surgical procedure of abdominoplasty for histological analysis. The reassessment will be carried out three times, being 30, 60 and 90 days after the initial session, with the repetition of all mentioned exams and photos for analysis of the results, of all participants.

DETAILED DESCRIPTION:
The search for efficient aesthetic treatments has been growing in a large part of the female public, among them the most common are body remodeling with a reduction in localized fat and improvement in the appearance of the skin when the individual has some degree of skin flaccidity.

Such unsightly conditions are characterized by intrinsic and extrinsic changes in the individual, with localized fat being associated with a disturbance between consumption, expenditure and supply of related nutrients, poor diet, sedentary lifestyle where triglycerides will be stored in excess in pre-dominant areas, and skin flaccidity characterized by the reduction of fibroblasts, compromising the activity of collagen and elastin proteins responsible for support and elasticity, which may be related to external factors such as pregnancy, weight loss, among others. For the treatment of these aesthetic affections, different treatment options emerged, both invasive and non-invasive.

Among the treatment options commonly used in dermatofunctional physiotherapy that can contribute to body remodeling and improvement in the appearance of the skin are ultrasound, carboxytherapy, shockwave therapy and radiofrequency, among others. Within the radiofrequency range is Tecartherapy, High Frequency Capacitive and Resistive Electrical Transfer Therapy which, however, is already known scientifically with good clinical and scientific results in orthopedic physiotherapy for the rehabilitation of muscle injuries. However, some researchers have proposed that the physiological effects of Tecartherapy may favor the treatment of various unsightly conditions, especially wrinkles and skin sagging, as well as the treatment of cellulite and localized fat.

According to authors, the heat generated by Tecartherapy acts on the fat cell and the extracellular matrix, in order to produce reversible and irreversible damage to the cells. This situation can lead to changes in the stability of the phospholipid membrane, which are usually followed by cell breakdown and lysis, lipolysis.

In the skin, Tecartherapy can favor the stimulation of the dermis by radiofrequency and induce an immediate retraction of collagen fibers and promote the activation of fibroblasts by a mild thermally mediated lesion that induces the synthesis of new collagen fibers (neocollagenesis) and elastic fibers ( neoelastogenesis).

Thus, given the possible physiological effects of Tecartherapy and the scarcity of studies on the effectiveness of the technology in the treatment of localized fat and skin sagging, this study is justified with the objective of investigating the effects of the technology, determining its clinical and histological results in these unsightly conditions.

ELIGIBILITY:
Inclusion Criteria:

* participants must be aged between 30 and 45 years of age.
* body mass index considered normal or overweight 18.5 to 29.9.
* sedentary.
* with fat located above 1.5cm and sagging abdominal skin.
* which cannot be under other aesthetic treatments for the same purpose.
* must have preserved local understanding and sensitivity.

Exclusion Criteria:

* participants who present alteration in sensitivity.
* who have contraindications for the use of the therapeutic resource used in the research, which are:
* Electronic device implanted as a cardiac pacemaker;
* Large metallic implant in the treated area;
* Pregnant patients;
* Patients with venous insufficiency of the lower limbs;
* About neoplastic areas;
* Osteoporosis;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical procedures | one month
  Immunohistochemical reactions were performed on 3μm-thick sections, arranged on silanized slides. The antibodies used were: polyclonal anti-Caspase3 , monoclonal anti-Cleaved Caspase 3 ; monoclonal anti-CD68, monoclonal anti-hormone-sensitive lipase - HSL - and Adipophilin. After preparing the slides, they were analyzed with a DMR microscope (Leica), and photographs were taken at 400x magnification. To quantify the analyses, the ImageJ® software (NIH, Bethesda, USA) was used.
  All reactions were performed following the manufacturers' protocol and all were standardized by the pathological analysis laboratory of the Hospital de Clínicas da Unicamp. The quantification of immunostaining was performed considering the number of positive cells and intensity, with final scores ranging from

CONTACTS AND LOCATIONS:
Locations (1):
- Ibramed - Indústria Brasileira de Equipamentos Médicos, Amparo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Contact the responsible researcher, we can provide the participant data